CLINICAL TRIAL: NCT05579210
Title: Developing and Implementing an Online Relapse Prevention Psychotherapy Program for Patients With Alcohol Use Disorder
Brief Title: Online Relapse Prevention Therapy for Patients With Alcohol Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Nazanin Alavi (Other)
Responsible Party: Sponsor-Investigator, Dr. Nazanin Alavi, Principal investigator, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6033212
Record Dates: First submitted 2022-10-07; First posted 2022-10-13 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either receive 10 weekly session of online relapse prevention therapy (e-RPT) or 10 weekly sessions of face-to-face relapse prevention therapy (RPT).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online relapse prevention therapy (eRPT) (Experimental): Online relapse preventiontherapy
  Interventions: Behavioral: Online relapse prevention therapy
- Face-to-face relapse prevention therapy (RPT) (Active Comparator): Face-to-face in-person relapse prevention therapy
  Interventions: Behavioral: Face to face relapse prevention therapy

INTERVENTIONS:
Behavioral: Online relapse prevention therapy — Participants in the e-RPT group will receive 10 weekly predesigned online modules. The content of this program will involve interactive therapy modules based on the principles of. On average each module consists of 30 slides and should take approximately 45 minutes to complete. At the end of each module, participants will be assigned homework to be completed and submitted to their respective therapists up to 48 hours before their next weekly session. The therapists will develop personalized feedback by using session-specific therapy feedback templates. These templates ensure that feedback is also more standardized and structured between different patients and therapists. In previous studies, therapists have been able to effectively use these templates to prepare feedback in approximately 15-20 minutes. The contents of each session are outlined on the detailed description section.
  Other Names: e-RPT
  Arms: Online relapse prevention therapy (eRPT)
Behavioral: Face to face relapse prevention therapy — Participants in the face-to-face intervention will meet with their therapist weekly through Microsoft Teams (video conference). During these 1-hour sessions, therapists will follow the same 10-week structure and content as e-RPT. Though compared to e-RPT, in face-to-face sessions, the homework will be reviewed with the participant, during the session, providing the appropriate feedback. Then the therapists will prepare a weekly patient report of each session for the principal investigator. At the end of each session, participants will receive the same homework as the e-RPT condition which they will receive feedback on during the following face-to-face session. Following the 10-week face-to-face intervention, participants will have the opportunity to join the e-RPT program.
  Other Names: RPT
  Arms: Face-to-face relapse prevention therapy (RPT)

SUMMARY:
Alcohol use disorder (AUD) is characterized by problematic alcohol use accompanied by clinically significant distress. This disorder is associated with high relapse rates, with one in five patients remaining abstinent 12 months post-treatment. Traditional face-to-face relapse prevention treatment (RPT) is a form of cognitive behavioural therapy that examines one's situational triggers, maladaptive thought processes, self-efficacy, and motivation, however access to this treatment is frequently limited due to its high cost, long waitlists, and inaccessibility. Thus, an online adaptation of RPT (e-RPT) could address these limitations by providing a more cost-effective and accessible delivery method for mental health care in this population. This study aims to establish the first academic e-RPT program to address AUD in the general population. We will recruit adult participants (n = 60) with a confirmed diagnosis of AUD. Then, these participants will be randomly assigned to receive ten sessions of e-RPT or face-to-face RPT. e-RPT will consist of 10 predesigned modules and homework with asynchronous personalized feedback from a therapist. Face-to-face RPT will consist of 10, one-hour long face-to-face sessions with a therapist. The predesigned modules and the face-to-face sessions will present the same content and structure. Self-efficacy, resilience, depressive symptomatology, and alcohol consumption will be measured through various questionnaires at baseline, week 5, and week 10. Outcome data will be assessed using linear and binomial regression (continuous and categorical outcomes respectively). Qualitative data will be analyzed using thematic analysis methods.

DETAILED DESCRIPTION:
Participants (n = 60) diagnosed with AUD will be recruited through physician referrals from Kingston Health Sciences Centre, family physicians, and other healthcare providers, and self-referrals in Kingston, Ontario. After providing consent to participate in the study, a Mini International Neuropsychiatric Interview 7.0.2 (MINI) will be conducted to confirm the diagnosis of mild to moderate AUD and other eligibility parameters (Sheehan et.al. 1981). The MINI is a diagnostic interview that assesses 17 common mental disorders by following the Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5) diagnostic criteria (Sheehan et.al. 1981). After the MINI, the Readiness To Change Questionnaire (RCQ) will be administered in an interview format to understand the individual's desire to change their alcohol consumption (Rollnick et.al. 1992). In addition to the RCQ, participants will be asked the following questions to get a better understanding of their history of AUD: Have you been diagnosed with AUD?; If Applicable: When were you diagnosed with AUD?; Are you currently enrolled in another relapse prevention program?; In the past month how many times have you had an alcoholic beverage?; If applicable: in those times, on average how many drinks did you have?; If applicable: in the past month on average, how many drinks did you have per week? The intake MINI and questions will be reviewed with the head psychiatrist, to ensure that the participant meets eligibility criteria and to confirm the diagnosis of AUD.

Interventions Upon completion of the eligibility assessments, participants will be randomly assigned through a computerized system to one of two groups; e-RPT or face-to-face RPT. Participants will be equally stratified (e-RPT n = 30; face-to-face RPT n = 30). These treatments will be delivered as an augmentation to treatment as usual (TAU) (e.g., medications, regular physician or clinician visits, referrals or consultations that are conducted outside of the current research study). The e-RPT program will be delivered through the Online Psychotherapy Tool (OPTT; OPTT Inc.), a secure and interactive platform developed by the Queen's Online Psychotherapy Lab (QUOPL). The face-to-face RPT program will be delivered through video conference sessions using Microsoft Teams. However, it is important to note that participants in the face-to-face group will also have access to OPTT. Participants in both groups will need access to OPTT to complete module 0 before starting with their respective programs, and to access their drinking diary to report their daily drinking. Module 0 will only serve to quickly introduce participants to OPTT, and the programs and to access their drinking diary.

E-RPT

Participants in the e-RPT group will receive 10 weekly predesigned online modules. The content of this program will involve interactive therapy modules and homework, for which participants will receive asynchronous individualized feedback from a therapist each week. Participants in the e-RPT condition will receive one module per week and have continuous access to them on the OPTT platform. On average each module consists of 30 slides and should take approximately 45 minutes to complete. At the end of each module, participants will be assigned homework to be completed and submitted to their respective therapists up to 48 hours before their next weekly session. The therapists will develop personalized feedback by using session-specific therapy feedback templates. These templates ensure that feedback is also more standardized and structured between different patients and therapists. In previous studies, therapists have been able to effectively use these templates to prepare feedback in approximately 15-20 minutes. Therefore, compared to one-hour-long face-to-face therapy sessions, online sessions require around 15-20 minutes of therapist time, which can enhance the scalability of the online intervention and increase the number of individuals assigned to a therapist. Following the principles of CBT and RPT, this e-RPT program will focus on teaching essential cognitive and behavioural skills such as identifying maladaptive thought processes, increasing engagement in day-to-day activities, and developing strategies to reduce alcohol consumption. The content of the sessions is outlined below:

* Session 1: Understanding Addiction - Introduces relapse prevention and what to expect from the course. The session explains what addiction is, including symptoms, signs, consequences, and the different types of addiction. Participants will create a SMART goal that they will try to achieve throughout the weeks. They will also share their personal experience with addiction
* Session 2: Exploring and Strengthening Your Motivation - Focuses on the five stages of motivation and the role of motivation in relapse prevention. Helpful techniques are discussed to reflect on and boost motivation throughout their recovery journey. Participants will create a pros and cons list about stopping alcohol use and will reflect on different aspects of their ability to stop using alcohol.
* Session 3: Triggers - Describes what triggers are and how to recognize them, including both internal and external triggers. This session also provides strategies for how to handle triggers through avoidance and careful planning. Participants will be asked to identify their triggers and how to prepare for them if encountered.
* Session 4: Handling Cravings and Signs of Relapse - Presents skills to use when confronting cravings, and how to identify and prevent a potential relapse. For instance, by applying distraction methods when they experience stressful situations to decrease their urge to consume alcohol. Also, it asks participants to identify their warning signs by reflecting on previous relapse experiences.
* Session 5: The 5-Part Model - Provides further introduction about CBT and its components. Also, it explains the 5 Part Model, which highlights the importance of differentiating between our thoughts, feelings, physical reactions, and behaviours in stressful situations. Participants are asked to complete the 5 Part Model with an example from their life.
* Session 6: The Thought Record - Part 1 - Introduces the thought record and its relation to CBT to help in the understanding of the connection between feelings, behaviours, and thoughts. This session focuses on the first three columns of the Thought Record (out of 7 columns). The first three columns include the situation, followed by the feelings and automatic thoughts associated with the situation. Participants are asked to complete the first three columns of a thought record for a stressful situation they experienced within the past week.
* Session 7: The Thought Record - Part 2 - This session continues with the remaining 4 columns of the Thought Record including, gathering evidence in support and against the identified automatic thoughts, and finding alternative and balanced thoughts after examining the evidence. Thus, this session highlights how to challenge irrational thoughts by developing more balanced and helpful thoughts. Participants have to complete a full thought record from a stressful situation related to their AUD within the past week.
* Session 8: Thinking Errors and The Activity Record - Explores irrational thinking and common thinking errors. This session also presents and highlights the importance of the Activity Record; a tool designed to record and plan weekly activities. Participants are asked to complete an activity record for an entire week.
* Session 9. Mindfulness and Breathing Techniques - Presents mindfulness, breathing techniques, and other helpful skills to reduce urges and cravings associated with alcohol and to promote increased awareness. Participants are asked to incorporate one or more of these practices into their daily routines for a week and to reflect on how these practices made them feel. Also, to reflect on which practice, if any, they found to be the most effective.
* Session 10. Review - This session is a review of the program. It summarizes all the useful tools and techniques for relapse prevention learned throughout the program. Participants are asked to reflect on the activities that they found to be the most effective throughout the sessions.

Face-to-Face RPT Participants in the face-to-face intervention will meet with their therapist weekly through Microsoft Teams (video conference). During these 1-hour sessions, therapists will follow the same 10-week structure and content as e-RPT. Though compared to e-RPT, in face-to-face sessions, the homework will be reviewed with the participant, during the session, providing the appropriate feedback. Then the therapists will prepare a weekly patient report of each session for the principal investigator. At the end of each session, participants will receive the same homework as the e-RPT condition which they will receive feedback on during the following face-to-face session. Following the 10-week face-to-face intervention, participants will have the opportunity to join the e-RPT program.

Training Therapists for both e-RPT and face-to-face RPT will consist of research assistants who are trained in RPT and writing feedback. All therapists are trained by the principal investigator, who is an expert in the electronic delivery of psychotherapy (Alavi and Hirji 2020, Alavi et.al. 2016, Alavi and Omrani 2018). During training, the principal investigator will closely guide the therapists through their first patient (assigning modules, reviewing homework, writing feedback, and conducting face-to-face sessions). Then through the study, the therapists will be supervised by the principal investigator to ensure the quality and reliability of the treatment programs. To ensure the quality of the feedback, therapists will practice by writing feedback on practice homework templates. All feedback will be examined and revised by the principal investigator before being sent to the participants.

Ethics and privacy All components of this study were approved by the Queen's University Health Sciences and Affiliated Teaching Hospitals Research Ethics Board (TRAQ: 6033212). Participants were only identifiable by an ID number and hard copies of consent forms were stored securely on-site and will be destroyed 5 years after study completion. Participant data was only accessible by the care providers and anonymized data was provided to the analysis team. Participants could withdraw from the study at any point and request for their data to be removed from the analysis. The research team will safeguard the privacy of the participants to the extent permitted by the applicable laws and duty to report. OPTT is Health Insurance Portability and Accountability Act, Personal Information Protection and Electronic Documents Act, and Service Organization Control - 2 compliant. All servers and databases are hosted in Amazon Web Service Canada cloud infrastructure to assure provincial and federal privacy and security regulations are met. OPTT does not collect identifiable personal information or IP addresses. OPTT collects anonymized metadata to improve service quality and provide advanced analytics to the clinician team.

Data Analysis At first, data will be assessed for outliers, missing, and/or nonsensical variables. These variables will not be imputed since they will be handled as missing. Similar studies that involved CBT and e-CBT demonstrated a drop-out rate of up to 40% for both conditions once the study concluded (Bados et.al. 2007). Thus, this study will intentionally over-sample the experimental and control groups to account for this drop-out rate. Given that several outcomes will be used, it is difficult to calculate a single sample size or provide a specific power calculation. However, applying the IMMPACT recommendations for treatment outcomes associated with pain and function, the minimal clinically important difference (MCID) for mood related outcomes is a change higher than 2 to 12 points in mood related scores from baseline (Dworkin et.al. 2008, Gatchel et.al. 2013). Thus, with a sample of 60 participants (30 per arm) and applying the sample size calculation presented by Rosner (2011) with p = 0.05 and a power of 0.95, our study would be able to significantly detect changes in mood scores of 3 to 12 points or higher (depending on the scale). Baseline mood scores related to AUD applied to the sample size calculation were obtained from the literature (O'Reilly et.al. 2019, Jordans et.al. 2019). Using Mann-Whitney-U tests, demographic information from individuals who completed the program and those who dropped out will be compared to identify possible differences. Additionally, an intention-to-treat analysis will be conducted to assess the clinical effects of the program on participants who dropped out prematurely. Linear regression (continuous outcomes) and binomial regression analysis (categorical outcomes) were used to identify variables associated with outcome measures. Comparative analysis between groups was analyzed using group and paired t-tests. OPTT collected usage statistics (i.e., number of logins per day, amount of time spent logged in) will be compared to face-to-face metrics to determine cost and time savings between the two programs.

Current progress According to the literature on the efficacy of CBT in AUD we hypothesize that both e-RPT and face-to-face RPT will reduce alcohol consumption, relapse(s) risk, and improve other outcome measures of interest (depressive symptom, self-efficacy, quality of life, and resilience) (Connor et.al. 2016). This randomized controlled trial was approved by the Queen's University Health Science and Affiliated Teaching Hospitals Research Ethics Board in April 2022 and began recruitment in October 2022. We expect to finalize recruitment and data gathering in October 2023 and analyze the findings by December 2023 at which point we will begin our process of knowledge dissemination (including but not limited to peer-reviewed publications, scientific presentations, grant proposals, and reports).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mild to moderate AUD according to the DSM-5
* Competence to consent to participate in the study
* Ability to speak and read English
* Consistent and reliable access to the internet
* In contemplation stage of change (according to Readiness for change questionnaire) related to stopping drinking or having stopped consuming alcohol in the past 30 days

Exclusion Criteria:

* Acute hypomanic/manic episodes
* Acute psychosis
* Active substance use disorder classified as moderate or severe according to the DSM-5
* Active suicidal or homicidal ideation
* Untreated clinically significant somatic symptoms or mental disorders (PHQ ≥ 15, GAD-7 ≥ 15)
* Current enrolment in another relapse prevention program
* Men who drink more than four drinks per day or 14 drinks per week and women who drink three drinks per day or seven drinks per week in the past month

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-04-23 (Actual); Study Completion 2024-04-23 (Actual)

PRIMARY OUTCOMES:
Change in daily drinking using a Drink diary | Daily records in drinking diary from baseline (week 0) to study endpoint (10 weeks)
  Records daily drinking in standard drinks, setting of drinks, if participant drank with someone else, and if the drinking resulted in hospitalization that day.

SECONDARY OUTCOMES:
Self-efficacy at resisting craving or urges to engage in addictive behaviour using the Situational Confidence Questionnaire (SCQ-100) | Baseline (pre treatment), week 5 (mid treatment), week 10 (post treatment)
  Self-efficacy will be measured through the Situational Confidence Questionnaire (SCQ-100) which is a self-report that consists of 100 items and 8 subscales [42]. The SCQ-100 examines experiences that people with AUD have concerning relapse or excessive drinking [42].
Quality of life changes from baseline using the Quality of Life Enjoyment and Satisfaction Questionnaire- Short Form (Q-LES-Q-SF) | Baseline (pre treatment), week 5 (mid treatment), week 10 (post treatment)
  Quality of life will be measured using the Quality of Life Enjoyment and Satisfaction Questionnaire- Short Form (Q-LES-Q-SF) [43]. This 16-item self-reported questionnaire explores topics related to health including a participant's leisure activities, medication satisfaction, mood, and physical health [43]. A five-point scale is used to assess different aspects of an individual's life. A score of 1 indicates that the specific part of the person's life is very poor and a score of 5 indicates that it is very good [43]
Resilience changes from baseline using the 14-item Resilience Scale (RS-14) | Baseline (pre treatment), week 5 (mid treatment), week 10 (post treatment)
  The 14-item Resilience Scale (RS-14) will be used to measure resilience [45]. The RS-14 presents 14 statements to the participant with responses ranging from 1 meaning they strongly disagree with the statement to 7 indicating that they strongly agree with the statement [45].
Coping behaviours and thoughts changes from baseline using the Coping Behaviors Inventory (CBI) | Baseline (pre treatment), week 5 (mid treatment), week 10 (post treatment)
  Behaviours and thoughts that can aid in preventing, avoiding, and controlling the resumption of heavy drinking will be measured through the Coping Behaviors Inventory (CBI) [47]. The CBI is a 36-item self-report questionnaire with two subscales of 14 cognitive and 22 behavioural questions [47]. This scale assesses various thoughts and behaviours that a person with AUD might use to decrease or avoid alcohol consumption [47].
Depressive Symptomatology changes from baseline using the Patient Health Questionnaire (PHQ-9) | Baseline (pre treatment), week 5 (mid treatment), week 10 (post treatment)
  Depressive Symptomatology will be measured through the Patient Health Questionnaire (PHQ-9) [48]. This 9-item self-report questionnaire assesses a participant's depressive symptomatology in the last two weeks [48]. Answers are measured on a scale of 0 meaning, not at all to 3 indicating that the person experiences the statement nearly every day [48]
Efficiency of therapist's time comparing time spent writing personalized feedback to time spent conducting the face-to-face sessions | Once a week for the 10 weeks of the program
  Involves determining whether using e-RPT is more time efficient than face-to-face RPT. Thus, this study will track the amount of time that e-RPT therapists spend writing feedback compared to the one-hour face-to-face session as a measure of therapists' time efficiency.

OTHER OUTCOMES:
Qualitative assessment of treatment engagement through the program, by looking at module completion, and adherence to the program | Once a week for the 10 weeks of the program
  Behavioural data regarding patients' interaction and engagement with their therapy such as module and homework completion in e-RPT, and session attendance in face-to-face RPT will be collected to provide qualitative information about these programs.

CONTACTS AND LOCATIONS:
Overall Officials: Nazanin Alavi, MD, Principal Investigator — Queen's University
Locations (1):
- Queen's University Online Psychotherapy lab, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
IPD won't be shared with other researchers

REFERENCES:
- [Background] Rehm J, Mathers C, Popova S, Thavorncharoensap M, Teerawattananon Y, Patra J. Global burden of disease and injury and economic cost attributable to alcohol use and alcohol-use disorders. Lancet. 2009 Jun 27;373(9682):2223-33. doi: 10.1016/S0140-6736(09)60746-7. PMID 19560604
- [Background] Grant BF, Stinson FS, Dawson DA, Chou SP, Dufour MC, Compton W, Pickering RP, Kaplan K. Prevalence and co-occurrence of substance use disorders and independent mood and anxiety disorders: results from the National Epidemiologic Survey on Alcohol and Related Conditions. Arch Gen Psychiatry. 2004 Aug;61(8):807-16. doi: 10.1001/archpsyc.61.8.807. PMID 15289279
- [Background] Kranzler HR, Soyka M. Diagnosis and Pharmacotherapy of Alcohol Use Disorder: A Review. JAMA. 2018 Aug 28;320(8):815-824. doi: 10.1001/jama.2018.11406. PMID 30167705
- [Background] Castillo-Carniglia A, Keyes KM, Hasin DS, Cerda M. Psychiatric comorbidities in alcohol use disorder. Lancet Psychiatry. 2019 Dec;6(12):1068-1080. doi: 10.1016/S2215-0366(19)30222-6. Epub 2019 Oct 17. PMID 31630984
- [Background] Rehm J. The risks associated with alcohol use and alcoholism. Alcohol Res Health. 2011;34(2):135-43. PMID 22330211
- [Background] Rosner B. Fundamentals of Biostatistics. 7th ed. Boston, MA: Brooks/Cole; 2011
- [Background] Samokhvalov AV, Popova S, Room R, Ramonas M, Rehm J. Disability associated with alcohol abuse and dependence. Alcohol Clin Exp Res. 2010 Nov;34(11):1871-8. doi: 10.1111/j.1530-0277.2010.01275.x. PMID 20662803
- [Background] World Health Organization. International classification of functioning, disability and health. 2001
- [Background] The Lancet Gastroenterology Hepatology. Drinking alone: COVID-19, lockdown, and alcohol-related harm. Lancet Gastroenterol Hepatol. 2020 Jul;5(7):625. doi: 10.1016/S2468-1253(20)30159-X. No abstract available. PMID 32553138
- [Background] Da BL, Im GY, Schiano TD. Coronavirus Disease 2019 Hangover: A Rising Tide of Alcohol Use Disorder and Alcohol-Associated Liver Disease. Hepatology. 2020 Sep;72(3):1102-1108. doi: 10.1002/hep.31307. PMID 32369624
- [Background] Tull MT, Edmonds KA, Scamaldo KM, Richmond JR, Rose JP, Gratz KL. Psychological Outcomes Associated with Stay-at-Home Orders and the Perceived Impact of COVID-19 on Daily Life. Psychiatry Res. 2020 Jul;289:113098. doi: 10.1016/j.psychres.2020.113098. Epub 2020 May 12. PMID 32434092
- [Background] Clay JM, Parker MO. Alcohol use and misuse during the COVID-19 pandemic: a potential public health crisis? Lancet Public Health. 2020 May;5(5):e259. doi: 10.1016/S2468-2667(20)30088-8. Epub 2020 Apr 8. No abstract available. PMID 32277874
- [Background] Kim JU, Majid A, Judge R, Crook P, Nathwani R, Selvapatt N, Lovendoski J, Manousou P, Thursz M, Dhar A, Lewis H, Vergis N, Lemoine M. Effect of COVID-19 lockdown on alcohol consumption in patients with pre-existing alcohol use disorder. Lancet Gastroenterol Hepatol. 2020 Oct;5(10):886-887. doi: 10.1016/S2468-1253(20)30251-X. Epub 2020 Aug 5. No abstract available. PMID 32763197
- [Background] Barrick C, Connors GJ. Relapse prevention and maintaining abstinence in older adults with alcohol-use disorders. Drugs Aging. 2002;19(8):583-94. doi: 10.2165/00002512-200219080-00004. PMID 12207552
- [Background] Sobell MB, Sobell LC. Controlled drinking after 25 years: how important was the great debate? Addiction. 1995 Sep;90(9):1149-53; discussion 1157-77. No abstract available. PMID 7580815
- [Background] Chick JD. Book Review: Alcoholism Treatment in Transition. 1981
- [Background] Hunt WA, Barnett LW, Branch LG. Relapse rates in addiction programs. J Clin Psychol. 1971 Oct;27(4):455-6. doi: 10.1002/1097-4679(197110)27:43.0.co;2-r. No abstract available. PMID 5115648
- [Background] Pearson FS, Prendergast ML, Podus D, Vazan P, Greenwell L, Hamilton Z. Meta-analyses of seven of the National Institute on Drug Abuse's principles of drug addiction treatment. J Subst Abuse Treat. 2012 Jul;43(1):1-11. doi: 10.1016/j.jsat.2011.10.005. Epub 2011 Nov 25. PMID 22119178
- [Background] Miller WR, Wilbourne PL. Mesa Grande: a methodological analysis of clinical trials of treatments for alcohol use disorders. Addiction. 2002 Mar;97(3):265-77. doi: 10.1046/j.1360-0443.2002.00019.x. PMID 11964100
- [Background] Carroll KM, Kiluk BD. Cognitive behavioral interventions for alcohol and drug use disorders: Through the stage model and back again. Psychol Addict Behav. 2017 Dec;31(8):847-861. doi: 10.1037/adb0000311. Epub 2017 Aug 31. PMID 28857574
- [Background] Monti, P. M., Kadden, R. M., Rohsenow, D. J., Cooney, N. L., & Abrams, D. B. (2002). (2nd ed.). Guilford Press.
- [Background] Heather N, Stockwell T. The Essential Handbook of Treatment and Prevention of Alcohol Problems. J. Wiley; 2004
- [Background] Carroll, K. M. (1996). Relapse prevention as a psychosocial treatment: A review of controlled clinical trials. Experimental and Clinical Psychopharmacology, 4(1), 46-54. https://doi.org/10.1037/1064-1297.4.1.46
- [Background] Irvin JE, Bowers CA, Dunn ME, Wang MC. Efficacy of relapse prevention: a meta-analytic review. J Consult Clin Psychol. 1999 Aug;67(4):563-70. doi: 10.1037//0022-006x.67.4.563. PMID 10450627
- [Background] McCrady BS. Alcohol use disorders and the Division 12 Task Force of the American Psychological Association. Psychol Addict Behav. 2000 Sep;14(3):267-76. PMID 10998952
- [Background] Magill M, Ray L, Kiluk B, Hoadley A, Bernstein M, Tonigan JS, Carroll K. A meta-analysis of cognitive-behavioral therapy for alcohol or other drug use disorders: Treatment efficacy by contrast condition. J Consult Clin Psychol. 2019 Dec;87(12):1093-1105. doi: 10.1037/ccp0000447. Epub 2019 Oct 10. PMID 31599606
- [Background] Sinha R. The role of stress in addiction relapse. Curr Psychiatry Rep. 2007 Oct;9(5):388-95. doi: 10.1007/s11920-007-0050-6. PMID 17915078
- [Background] Probst C, Manthey J, Martinez A, Rehm J. Alcohol use disorder severity and reported reasons not to seek treatment: a cross-sectional study in European primary care practices. Subst Abuse Treat Prev Policy. 2015 Aug 12;10:32. doi: 10.1186/s13011-015-0028-z. PMID 26264215
- [Background] Johansson M, Sinadinovic K, Gajecki M, Lindner P, Berman AH, Hermansson U, Andreasson S. Internet-based therapy versus face-to-face therapy for alcohol use disorder, a randomized controlled non-inferiority trial. Addiction. 2021 May;116(5):1088-1100. doi: 10.1111/add.15270. Epub 2020 Oct 13. PMID 32969541
- [Background] Andersson G, Titov N. Advantages and limitations of Internet-based interventions for common mental disorders. World Psychiatry. 2014 Feb;13(1):4-11. doi: 10.1002/wps.20083. PMID 24497236
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Rollnick S, Heather N, Gold R, Hall W. Development of a short 'readiness to change' questionnaire for use in brief, opportunistic interventions among excessive drinkers. Br J Addict. 1992 May;87(5):743-54. doi: 10.1111/j.1360-0443.1992.tb02720.x. PMID 1591525
- [Background] Cougle JR, Summers BJ, Allan NP, Dillon KH, Smith HL, Okey SA, Harvey AM. Hostile interpretation training for individuals with alcohol use disorder and elevated trait anger: A controlled trial of a web-based intervention. Behav Res Ther. 2017 Dec;99:57-66. doi: 10.1016/j.brat.2017.09.004. Epub 2017 Sep 19. PMID 28941810
- [Background] Witkiewitz K, Stein ER, Votaw VR, Wilson AD, Roos CR, Gallegos SJ, Clark VP, Claus ED. Mindfulness-Based Relapse Prevention and Transcranial Direct Current Stimulation to Reduce Heavy Drinking: A Double-Blind Sham-Controlled Randomized Trial. Alcohol Clin Exp Res. 2019 Jun;43(6):1296-1307. doi: 10.1111/acer.14053. Epub 2019 May 9. PMID 30977904
- [Background] Dawson DA, Grant BF, Li TK. Quantifying the risks associated with exceeding recommended drinking limits. Alcohol Clin Exp Res. 2005 May;29(5):902-8. doi: 10.1097/01.alc.0000164544.45746.a7. PMID 15897737
- [Background] Drinking levels defined. National Institute on Alcohol Abuse and Alcoholism. https://www.niaaa.nih.gov/alcohol-health/overview-alcohol-consumption/moderate-binge-drinking.
- [Background] Fernandez E, Woldgabreal Y, Day A, Pham T, Gleich B, Aboujaoude E. Live psychotherapy by video versus in-person: A meta-analysis of efficacy and its relationship to types and targets of treatment. Clin Psychol Psychother. 2021 Nov;28(6):1535-1549. doi: 10.1002/cpp.2594. Epub 2021 May 5. PMID 33826190
- [Background] Alavi N, Hirji A. The Efficacy of PowerPoint-based CBT Delivered Through Email: Breaking the Barriers to Treatment for Generalized Anxiety Disorder. J Psychiatr Pract. 2020 Mar;26(2):89-100. doi: 10.1097/PRA.0000000000000455. PMID 32134882
- [Background] Alavi N, Hirji A, Sutton C, Naeem F. Online CBT Is Effective in Overcoming Cultural and Language Barriers in Patients With Depression. J Psychiatr Pract. 2016 Jan;22(1):2-8. doi: 10.1097/PRA.0000000000000119. PMID 26813483
- [Background] Alavi N, Yang M, Stephenson C, Nikjoo N, Malakouti N, Layzell G, Jagayat J, Shirazi A, Groll D, Omrani M, O'Riordan A, Khalid-Khan S, Freire R, Brietzke E, Gomes FA, Milev R, Soares CN. Using the Online Psychotherapy Tool to Address Mental Health Problems in the Context of the COVID-19 Pandemic: Protocol for an Electronically Delivered Cognitive Behavioral Therapy Program. JMIR Res Protoc. 2020 Dec 18;9(12):e24913. doi: 10.2196/24913. PMID 33290245
- [Background] Baltieri DA, Daro FR, Ribeiro PL, de Andrade AG. Comparing topiramate with naltrexone in the treatment of alcohol dependence. Addiction. 2008 Dec;103(12):2035-44. doi: 10.1111/j.1360-0443.2008.02355.x. Epub 2008 Oct 8. PMID 18855810
- [Background] Low-risk alcohol drinking guidelines. Canada.ca. https://www.canada.ca/en/health-canada/services/substance-use/alcohol/low-risk-alcohol-drinking-guidelines.html. Published July 5, 2021
- [Background] Miller PJ, Ross SM, Emmerson RY, Todt EH. Self-efficacy in alcoholics: clinical validation of the Situational Confidence Questionnaire. Addict Behav. 1989;14(2):217-24. doi: 10.1016/0306-4603(89)90052-x. PMID 2728959
- [Background] Endicott J, Nee J, Harrison W, Blumenthal R. Quality of Life Enjoyment and Satisfaction Questionnaire: a new measure. Psychopharmacol Bull. 1993;29(2):321-6. PMID 8290681
- [Background] Stevanovic D. Quality of Life Enjoyment and Satisfaction Questionnaire-short form for quality of life assessments in clinical practice: a psychometric study. J Psychiatr Ment Health Nurs. 2011 Oct;18(8):744-50. doi: 10.1111/j.1365-2850.2011.01735.x. Epub 2011 May 5. PMID 21896118
- [Background] Aiena BJ, Baczwaski BJ, Schulenberg SE, Buchanan EM. Measuring resilience with the RS-14: a tale of two samples. J Pers Assess. 2015;97(3):291-300. doi: 10.1080/00223891.2014.951445. Epub 2014 Sep 25. PMID 25257682
- [Background] Zelviene P, Jovarauskaite L, Truskauskaite-Kuneviciene I. The Psychometric Properties of the Resilience Scale (RS-14) in Lithuanian Adolescents. Front Psychol. 2021 May 21;12:667285. doi: 10.3389/fpsyg.2021.667285. eCollection 2021. PMID 34093364
- [Background] Litman GK, Stapleton J, Oppenheim AN, Peleg M. An instrument for measuring coping behaviours in hospitalized alcoholics: implications for relapse prevention treatment. Br J Addict. 1983 Sep;78(3):269-76. doi: 10.1111/j.1360-0443.1983.tb02511.x. No abstract available. PMID 6578829
- [Background] Lowe B, Unutzer J, Callahan CM, Perkins AJ, Kroenke K. Monitoring depression treatment outcomes with the patient health questionnaire-9. Med Care. 2004 Dec;42(12):1194-201. doi: 10.1097/00005650-200412000-00006. PMID 15550799
- [Background] Zuithoff NP, Vergouwe Y, King M, Nazareth I, van Wezep MJ, Moons KG, Geerlings MI. The Patient Health Questionnaire-9 for detection of major depressive disorder in primary care: consequences of current thresholds in a crosssectional study. BMC Fam Pract. 2010 Dec 13;11:98. doi: 10.1186/1471-2296-11-98. PMID 21144018
- [Background] Bados A, Balaguer G, Saldana C. The efficacy of cognitive-behavioral therapy and the problem of drop-out. J Clin Psychol. 2007 Jun;63(6):585-92. doi: 10.1002/jclp.20368. PMID 17457848
- [Background] Connor JP, Haber PS, Hall WD. Alcohol use disorders. Lancet. 2016 Mar 5;387(10022):988-998. doi: 10.1016/S0140-6736(15)00122-1. Epub 2015 Sep 3. PMID 26343838
- [Background] Andrews G, Davies M, Titov N. Effectiveness randomized controlled trial of face to face versus Internet cognitive behaviour therapy for social phobia. Aust N Z J Psychiatry. 2011 Apr;45(4):337-40. doi: 10.3109/00048674.2010.538840. Epub 2011 Feb 16. PMID 21323490
- [Background] Coates JM, Gullo MJ, Feeney GFX, Young RM, Dingle GA, Connor JP. Alcohol expectancies pre-and post-alcohol use disorder treatment: Clinical implications. Addict Behav. 2018 May;80:142-149. doi: 10.1016/j.addbeh.2018.01.029. Epub 2018 Jan 31. PMID 29407685
- [Background] Sharma A, Das K, Sharma S, Ghosh A. Feasibility and preliminary effectiveness of internet-mediated 'relapse prevention therapy' for patients with alcohol use disorder: A pilot study. Drug Alcohol Rev. 2022 Mar;41(3):641-645. doi: 10.1111/dar.13395. Epub 2021 Oct 27. PMID 34704318
- [Background] Dworkin RH, Turk DC, Wyrwich KW, Beaton D, Cleeland CS, Farrar JT, Haythornthwaite JA, Jensen MP, Kerns RD, Ader DN, Brandenburg N, Burke LB, Cella D, Chandler J, Cowan P, Dimitrova R, Dionne R, Hertz S, Jadad AR, Katz NP, Kehlet H, Kramer LD, Manning DC, McCormick C, McDermott MP, McQuay HJ, Patel S, Porter L, Quessy S, Rappaport BA, Rauschkolb C, Revicki DA, Rothman M, Schmader KE, Stacey BR, Stauffer JW, von Stein T, White RE, Witter J, Zavisic S. Interpreting the clinical importance of treatment outcomes in chronic pain clinical trials: IMMPACT recommendations. J Pain. 2008 Feb;9(2):105-21. doi: 10.1016/j.jpain.2007.09.005. Epub 2007 Dec 11. PMID 18055266
- [Background] Gatchel RJ, Mayer TG, Choi Y, Chou R. Validation of a consensus-based minimal clinically important difference (MCID) threshold using an objective functional external anchor. Spine J. 2013 Aug;13(8):889-93. doi: 10.1016/j.spinee.2013.02.015. Epub 2013 Mar 21. PMID 23523434
- [Background] O'Reilly H, Hagerty A, O'Donnell S, Farrell A, Hartnett D, Murphy E, Kehoe E, Agyapong V, McLoughlin DM, Farren C. Alcohol Use Disorder and Comorbid Depression: A Randomized Controlled Trial Investigating the Effectiveness of Supportive Text Messages in Aiding Recovery. Alcohol Alcohol. 2019 Jan 9;54(5):551-558. doi: 10.1093/alcalc/agz060. PMID 31361815
- [Background] Jordans MJD, Luitel NP, Garman E, Kohrt BA, Rathod SD, Shrestha P, Komproe IH, Lund C, Patel V. Effectiveness of psychological treatments for depression and alcohol use disorder delivered by community-based counsellors: two pragmatic randomised controlled trials within primary healthcare in Nepal. Br J Psychiatry. 2019 Aug;215(2):485-493. doi: 10.1192/bjp.2018.300. Epub 2019 Jan 25. PMID 30678744
- [Derived] Eadie J, Gutierrez G, Moghimi E, Stephenson C, Khalafi P, Nikjoo N, Jagayat J, Gizzarelli T, Reshetukha T, Omrani M, Yang M, Alavi N. Developing and Implementing a Web-Based Relapse Prevention Psychotherapy Program for Patients With Alcohol Use Disorder: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2023 Jan 25;12:e44694. doi: 10.2196/44694. PMID 36567076

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-06): https://cdn.clinicaltrials.gov/large-docs/10/NCT05579210/Prot_SAP_000.pdf
  • Informed Consent Form (2022-10-06): https://cdn.clinicaltrials.gov/large-docs/10/NCT05579210/ICF_001.pdf